CLINICAL TRIAL: NCT04170296
Title: A Real World, Multicenter, Open-Label, Multiple Dose Study to Assess the Effectiveness of, and Satisfaction With, CCH Treatment of Buttocks or Thigh Cellulite in Adult Females
Brief Title: Real World CCH Study in Adult Females With Cellulite
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN3835-305
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Results first posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-01

CONDITIONS: Edematous Fibrosclerotic Panniculopathy (EFP); Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Posterolateral Thigh (Experimental): EN3835 up to 1.68mg (Collagenase Clostridium Histolyticum)
  Interventions: Drug: EN3835
- Cohort 2: Buttocks (Experimental): EN3835 up to 1.68mg (Collagenase Clostridium Histolyticum)
  Interventions: Drug: EN3835

INTERVENTIONS:
Drug: EN3835 — Collagenase Clostridium Histolyticum (CCH)

SUMMARY:
This is a multicenter, open-label, multiple dose, 2 cohort, Phase 3b study to assess the safety and efficacy of CCH in adult women with mild or moderate edematous fibrosclerotic panniculopathy (EFP).

Cohort 1 will include approximately 80 subjects with mild or moderate EFP in the posterolateral thighs and Cohort 2 will include approximately 70 subjects with mild or moderate EFP in the buttocks.

ELIGIBILITY:
Inclusion Criteria:

1. Have both buttocks or both posterolateral thighs with:

   1. A score of 2 or 3 (mild or moderate) as reported by the investigator using the Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS).
   2. A Hexsel Cellulite Severity Scale (CSS) Subsection D "Grade of Laxity, Flaccidity, or Sagging Skin" score of 0 (absence of laxity, flaccidity, or sagging skin), or 1 (slightly draped appearance) at the Screening Visit only.
2. Be willing to apply sunscreen to the treatment areas before each exposure to the sun for the duration of the study.
3. Be judged to be in good health.
4. Have a negative pregnancy test.
5. Be willing and able to cooperate with the requirements of the study.

Exclusion Criteria:

1. Is from a vulnerable population, as defined by the United States (US) Code of Federal Regulations (CFR) Title 45, Part 46, Section 46.111(b) and other local and national regulations, including but not limited to, employees (temporary, part-time, full-time, etc.) or a family member of the research staff conducting the study, or of the sponsor, or of the contract research organization, or of the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
2. Has a history of sensitivity or allergy to collagenase or any other excipient of CCH.
3. Has systemic conditions (coagulation disorders, malignancy, keloidal scarring, abnormal wound healing) that restricts study participation.
4. Has local (in areas to be treated) conditions (thrombosis, vascular disorder, active infection/inflammation, active cutaneous alteration, tattoo/mole) that restricts study participation.
5. Has skin laxity or linear undulations on the treatment region (both buttocks or both thighs) that can be effaced by lifting skin.
6. Has a Hexsel CSS Subsection D "Grade of laxity, flaccidity, or sagging skin" of 2 (moderate draped appearance) or 3 (severe draped appearance).
7. Requires anticoagulant or antiplatelet medication during the study.
8. Has used or intends to use any of the local applications/therapies/injections/procedures that restricts study participation.
9. Has received any collagenase treatments at any time prior to treatment in this study and/or has received previous treatment with EN3835 or CCH for cellulite.
10. Has received treatment with an investigational product within 30 days (or 5 half-lives, whichever is longer) of the Screening Visit.
11. Is pregnant and/or is providing breast milk in any manner, or plans to become pregnant and/or to provide breast milk during the course of the study.
12. Has any other condition(s) that, in the investigator's opinion, might indicate the subject to be unsuitable for the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 153 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2021-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hernandez, Study Director — Endo Pharmaceuticals
Locations (12):
- United States (11):
  - Endo Clinical Trial Site #2, Encino, California
  - Endo Clinical Trial Site #4, San Diego, California
  - Endo Clinical Trial Site #5, Solana Beach, California
  - Endo Clinical Trial Site #9, Westport, Connecticut
  - Endo Clinical Trial Site #1, Coral Gables, Florida
  - Endo Clinical Trial Site #10, Alpharetta, Georgia
  - Endo Clinical Trial Site #3, Chicago, Illinois
  - Endo Clinical Trial Site #11, Itasca, Illinois
  - Endo Clinical Trial Site #8, New Orleans, Louisiana
  - Endo Clinical Trial Site #6, New York, New York
  - Endo Clinical Trial Site #12, Nashville, Tennessee
- Endo Clinical Trial Site #7, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: Posterolateral Thigh | Cohort 2: Buttocks
Started | 81 | 72
Completed | 73 | 68
Not Completed | 8 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population includes all participants who have at least 1 injection of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Posterolateral Thigh | Cohort 2: Buttocks | Total
Number analyzed (Participants) | 81 | 72 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (9.40) | 42.7 (9.35) | 43.0 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 72 | 153
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 18 | 28
  Not Hispanic or Latino | 71 | 54 | 125
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 2 | 4
  White | 74 | 65 | 139
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 2 | 4
Weight [Mean (Standard Deviation); unit: kg] | 65.082 (8.3341) | 65.042 (8.9403) | 65.063 (8.5961)
Height [Mean (Standard Deviation); unit: cm] | 164.548 (6.2671) | 165.192 (6.6315) | 164.851 (6.4279)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.03 (2.640) | 23.89 (2.759) | 23.96 (2.689)
Skin Category (Fitzpatrick Scale) [Count of Participants; unit: Participants]
  I (Pale White) | 2 | 1 | 3
  II (Fair) | 33 | 24 | 57
  III (Darker White) | 24 | 28 | 52
  IV (Light Brown) | 18 | 14 | 32
  V (Brown) | 4 | 4 | 8
  VI (Dark Brown or Black) | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants With Improved (+1 or Better) Score on I-GAIS for Either Posterolateral Thigh
Description: Investigator Global Aesthetic Improvement Scale (I-GAIS) is a 7-point scale rating global aesthetic improvement in appearance, compared to pretreatment, as judged by the investigator. The rating categories are "Very Much Worse", "Much Worse", "Worse", "No Change", "Improved", "Much Improved", and "Very Much Improved".
Time Frame: 90 Days
Population: Evaluable Population includes all participants who have at least 1 injection of study medication and have at least 1 I-GAIS evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Posterolateral Thigh
Number analyzed (Participants) | 63
Participants | 58

2. Primary Outcome: The Proportion of Participants With Improved (+1 or Better) Score on I-GAIS for Either Buttock
Description: as for outcome 1
Time Frame: 90 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Buttocks
Number analyzed (Participants) | 61
Participants | 58

3. Secondary Outcome: Mean Change From Baseline in CR-PCSS for Each Buttock
Description: Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) is a 5-point photonumeric scale rating cellulite severity from "0" (none) to "4" (severe) from a clinician's perspective.
Time Frame: Day 22, 43, 90 and 180
Population: Evaluable Population includes all participants who received at least 1 injection of study medication and had at least 1 I-GAIS evaluation. Number of participants analyzed are evaluable population participants that had a change from baseline at the specified visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cohort 2: Buttocks (Left); Cohort 2: Buttocks (Right): EN3835 up to 1.68mg (Collagenase Clostridium Histolyticum)
  EN3835: Collagenase Clostridium Histolyticum (CCH)
Arm/Group | Cohort 2: Buttocks (Left) | Cohort 2: Buttocks (Right)
Number analyzed (Participants) | 71 | 71
units on a scale
  Day 22: number analyzed (Participants) | 69 | 69
  Day 22 | -0.3 (0.52) | -0.3 (0.50)
  Day 43: number analyzed (Participants) | 67 | 67
  Day 43 | -0.6 (0.63) | -0.5 (0.59)
  Day 90: number analyzed (Participants) | 61 | 61
  Day 90 | -0.7 (0.70) | -0.7 (0.53)
  Day 180: number analyzed (Participants) | 66 | 66
  Day 180 | -0.7 (0.63) | -0.6 (0.63)

4. Secondary Outcome: Mean Change From Baseline in Body Q Appraisal of Cellulite for Posterolateral Thigh Based on Total Score
Description: The Body-Q Appraisal of Cellulite is a subset of questions from the Body-Q questionnaire developed to measure participant perceptions of weight loss and/or body contouring. The minimum possible score is 11 and the maximum possible score is 44. Higher scores indicate the individual is less bothered by their cellulite. Copyright Memorial Sloan-Kettering Cancer Center
Time Frame: Day 90, Day 180
Population: Evaluable Population includes all participants who received at least 1 injection of study medication and had at least 1 I-GAIS evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: Posterolateral Thigh
Number analyzed (Participants) | 76
units on a scale
  Day 90: number analyzed (Participants) | 63
  Day 90 | 10.9 (9.84)
  Day 180: number analyzed (Participants) | 68
  Day 180 | 10.9 (9.76)

5. Secondary Outcome: Mean Change From Baseline in Body Q Appraisal of Cellulite for Buttock Based on Total Score
Description: as for outcome 4
Time Frame: Day 90, Day 180
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 2: Buttocks
Number analyzed (Participants) | 71
units on a scale
  Day 90: number analyzed (Participants) | 61
  Day 90 | 8.8 (8.38)
  Day 180: number analyzed (Participants) | 66
  Day 180 | 8.8 (9.57)

6. Secondary Outcome: The Proportion of Participants With Improved (+1 or Better) Score on I GAIS for Either Posterolateral Thigh
Description: as for outcome 1
Time Frame: Day 22, 43, and 180
Population: Population includes all participants who received at least 1 injection of study medication and had at least 1 I-GAIS evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Posterolateral Thigh
Number analyzed (Participants) | 76
Participants
  Day 22: number analyzed (Participants) | 70
  Day 22 | 64
  Day 43: number analyzed (Participants) | 67
  Day 43 | 59
  Day 180: number analyzed (Participants) | 68
  Day 180 | 61

7. Secondary Outcome: The Proportion of Participants With Improved (+1 or Better) Score on I-GAIS for Either Buttock
Description: as for outcome 1
Time Frame: Day 22, 43, and 180
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Buttocks
Number analyzed (Participants) | 71
Participants
  Day 22: number analyzed (Participants) | 69
  Day 22 | 50
  Day 43: number analyzed (Participants) | 67
  Day 43 | 62
  Day 180: number analyzed (Participants) | 66
  Day 180 | 59

8. Secondary Outcome: Percentage of Participants With Positive Antibody Titers for Anti-AUX-I and Anti AUX-II (Posterolateral Thigh)
Description: Immunogenicity samples with a positive titer value will undergo a log transformation for analyses. Samples with titer level less than 10 were assigned or imputed as a log transformed titer of 1 for analyses
Time Frame: Day 1, 90, and 180
Population: Safety Population includes all participants who received at least 1 injection of study medication
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Posterolateral Thigh (Anti AUX-I); Cohort 1: Posterolateral Thigh (Anti AUX-II): EN3835 up to 1.68mg (Collagenase Clostridium Histolyticum)
  EN3835: Collagenase Clostridium Histolyticum (CCH)
Arm/Group | Cohort 1: Posterolateral Thigh (Anti AUX-I) | Cohort 1: Posterolateral Thigh (Anti AUX-II)
Number analyzed (Participants) | 81 | 81
Participants
  Day 1 | 5 | 5
  Day 90: number analyzed (Participants) | 60 | 60
  Day 90 | 60 | 60
  Day 180: number analyzed (Participants) | 68 | 68
  Day 180 | 68 | 68

9. Secondary Outcome: Percentage of Participants With Positive Antibody Titers for Anti-AUX-I and Anti AUX-II (Buttocks)
Description: as for outcome 8
Time Frame: Day 1, 90 and 180
Population: Safety Population includes all participants who received at least 1 injection of study medication
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Buttocks (Anti AUX-I); Cohort 2: Buttocks (Anti AUX-II): EN3835 up to 1.68mg (Collagenase Clostridium Histolyticum)
  EN3835: Collagenase Clostridium Histolyticum (CCH)
Arm/Group | Cohort 2: Buttocks (Anti AUX-I) | Cohort 2: Buttocks (Anti AUX-II)
Number analyzed (Participants) | 72 | 72
Participants
  Day 1 | 7 | 5
  Day 90: number analyzed (Participants) | 61 | 61
  Day 90 | 61 | 61
  Day 180: number analyzed (Participants) | 66 | 66
  Day 180 | 66 | 65

10. Secondary Outcome: Presence of Neutralizing Antibody (NAb) Anti AUX-I and AUX-II (Posterolateral Thigh)
Description: All the samples with positive ADAs for the participants who had had every other titer levels in the first quartile and fourth quartile of all positive ADAs at Day 90 (performed separately for AUX-I and AUX-II) were tested for NAb.
Time Frame: Day 1, 90 and 180
Population: Subset of Safety Population samples were analyzed for NAbs. All the samples with positive ADAs for the participants who had had every other titer levels in the first quartile and fourth quartile of all positive ADAs at Day 90 (performed separately for AUX-I and AUX-II) were tested for NAb. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for the assessment. Percentages are based on number of participants tested for NAb at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Posterolateral Thigh (Anti AUX-I) | Cohort 1: Posterolateral Thigh (Anti AUX-II)
Number analyzed (Participants) | 13 | 17
Participants
  Day 1: number analyzed (Participants) | 2 | 1
  Day 1: Positive | 1 | 0
  Day 1: Negative | 1 | 1
  Day 90: Positive | 13 | 16
  Day 90: Negative | 0 | 1
  Day 180: number analyzed (Participants) | 11 | 15
  Day 180: Positive | 8 | 12
  Day 180: Negative | 3 | 3

11. Secondary Outcome: Presence of NAb Anti AUX-I and AUX-II (Buttocks)
Description: as for outcome 10
Time Frame: Day 1, 90 and 180
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Buttocks (Anti AUX-I) | Cohort 2: Buttocks (Anti AUX-II)
Number analyzed (Participants) | 17 | 13
Participants
  Day 1: number analyzed (Participants) | 2 | 2
  Day 1: Positive | 2 | 2
  Day 1: Negative | 0 | 0
  Day 90: Positive | 15 | 9
  Day 90: Negative | 2 | 4
  Day 180: Positive | 15 | 9
  Day 180: Negative | 2 | 4

ADVERSE EVENTS:
Time Frame: Time of informed consent signature until Day 180
Description: All serious and non-serious AEs, whether elicited or observed during study visit or spontaneously reported by the participant, including events that occurred from the time the participant signed the study specific consent form until completion of or discharge from the study
Arm/Group | Cohort 1: Posterolateral Thigh | Cohort 2: Buttocks
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/72
Other Adverse Events (participants affected / at risk) | 75/81 | 69/72
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Posterolateral Thigh (N=81) | Cohort 2: Buttocks (N=72)
Injection site bruising (General disorders) | 70 (311) | 67 (327)
Injection site dermatitis (General disorders) | 0 (0) | 1 (1)
Injection site discolouration (General disorders) | 14 (32) | 24 (46)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 3 (18) | 2 (12)
Injection site mass (General disorders) | 4 (7) | 5 (10)
Injection site nodule (General disorders) | 7 (17) | 5 (14)
Injection site oedema (General disorders) | 8 (34) | 5 (22)
Injection site pain (General disorders) | 53 (244) | 57 (298)
Injection site pruritus (General disorders) | 10 (37) | 14 (35)
Injection site rash (General disorders) | 1 (2) | 0 (0)
Injection site reaction (General disorders) | 2 (3) | 0 (0)
Injection site swelling (General disorders) | 12 (32) | 13 (34)
Injection site warmth (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0)
Oral herpes (Infections and infestations) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood sodium increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Coronavirus test positive (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Nitrite urine present (Investigations) | 0 (0) | 1 (1)
Urine ketone body present (Investigations) | 1 (1) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Post-inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 5 (10) | 2 (4)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT04170296/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT04170296/SAP_001.pdf